CLINICAL TRIAL: NCT00819884
Title: A Randomised, Two Way Cross-Over, Single-Blind, Phase I Study to Evaluate 24-hr Glucose Profiles in Patients With T2DM When Dosed OD and BD on Top of Metformin for Four Days With AZD1656
Brief Title: To Evaluate 24-hr Glucose After OD vs BD AZD1656
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Klas Malmberg, MD, PhD, Prof. Medical Science Director, Emerging Products, AstraZeneca Pharmaceuticals
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: D1020C00017
Record Dates: First submitted 2009-01-08; First posted 2009-01-09 (Estimated); Last update posted 2009-05-07 (Estimated); Status verified 2009-05

CONDITIONS: Type II Diabetes
Keywords: Type II Diabetes; 24 hour glucose profile
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — AZD1656

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- 1 (Experimental): twice daily during 4 days
  Interventions: Drug: AZD1656
- 2 (Experimental): once daily during 4 days
  Interventions: Drug: AZD1656

INTERVENTIONS:
Drug: AZD1656 — Oral suspension

SUMMARY:
The purpose of this study is to compare the 24-hour glucose profiles in diabetic patients treated with metformin following once daily and twice daily oral dosing

ELIGIBILITY:
Inclusion Criteria:

* type II diabetes patients, female with non child-bearing potential
* Type 2 Diabetes Mellitus (T2DM) diagnosis confirmed by C-peptide >0.3nmol/L and no Glutamic acid decarboxylase (GAD) antibodies at enrolment (screening)
* Treatment with metformin as single therapy for T2DM for at least 30 days prior to enrolment and the metformin dose must have been unchanged during this period

Exclusion Criteria:

* History of ischemic heart disease, symptomatic heart failure, stroke, transitory ischemic attack or symptomatic peripheral vascular disease
* Any clinically significant abnormality identified on physical examination, laboratory test or ECG, which in the judgement of investigator would compromise the subject's safety or successful participation in the clinical study

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2009-01; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
24-hr glucose (Calculated plasma glucose AUC0-24, change in fasting plasma glucose) | Repeated sampling during the 24 hour period on day -1, 4 and 8

SECONDARY OUTCOMES:
Safety and tolerability (Adverse events (AEs) during the study, blood pressure (BP), pulse rate, safety laboratory variables (incl. glucose) and investigator's interpretation of electrocardiogram (ECG) | Frequent measurements during the study period
Pharmacokinetic variables (Area under the plasma conc vs. time curve (AUC0-24), maximum plasma conc (Cmax), time to reach maximum plasma conc(tmax), terminal elimination half-life and apparent oral clearance | Repeated sampling at pre-specified timepoints on day 4 and 8
Pharmacodynamics (S-Insulin AUC0-24 and C-peptide AUC0-24) | Repeated sampling during the 24 hour period on day -1, 4 and 8

CONTACTS AND LOCATIONS:
Overall Officials: Klas Malmberg, MD, PhD, Prof.,, Study Director — AstraZeneca R&D Mölndal; Emanuel P DeNoia, M.D, Principal Investigator — Healthcare Discoveries LLC Icon Development Solutions
Locations (1):
- Research Site, San Antonio, Texas, United States